CLINICAL TRIAL: NCT03276533
Title: Effects of Intravenous Dexmedetomidine, Lidocaine and Their Combination on Postoperative Inflammation Cytokines After Laparoscopic Hysterectomy With General Anesthesia
Brief Title: Dexmedetomidine Combined With Lidocaine Infusion Affect Inflammation Cytokines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Xu Siqi, Principal Investigator,Department of Anesthesiology, Anqing Municipal Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: xuzhang2013
Record Dates: First submitted 2017-08-23; First posted 2017-09-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia; Reaction
Keywords: dexmedetomidine; lidocaine; cytokine
MeSH Terms: interventions — Sodium Chloride; Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intravenous saline, dexmedetomidine and lidocaine (Experimental)
  Interventions: Drug: Saline; Drug: Lidocaine; Drug: Dexmedetomidine; Drug: Lidocaine plus Dexmedetomidine
- Intravenous saline, dexmedetomidine, lidocaine and combination (Experimental)
  Interventions: Drug: Saline; Drug: Lidocaine; Drug: Dexmedetomidine; Drug: Lidocaine plus Dexmedetomidine
- Intravenous saline,dexmedetomidine plus lidocaine (Experimental)
  Interventions: Drug: Saline; Drug: Lidocaine; Drug: Dexmedetomidine; Drug: Lidocaine plus Dexmedetomidine
- Intravenous saline, dexmedetomidine combined with lidocaine (Experimental)
  Interventions: Drug: Saline; Drug: Lidocaine; Drug: Dexmedetomidine; Drug: Lidocaine plus Dexmedetomidine

INTERVENTIONS:
Drug: Saline — Participants in the group CON were received normal saline infusion until 30 min before the end of the operation.Interleukin-6 and tumor necrosis factor-α levels in serum were measured at different time points: before administration of drugs (T1), at the end of the operation (T2), postoperative 2 hour (T3) and postoperative 24 hour (T4)
Drug: Lidocaine — Participants in the group LIDO received lidocaine infusion (1.5 mg/kg loading, 1.5 mg/kg/h infusion)until 30 min before the end of the operation.Interleukin-6 and tumor necrosis factor-α levels in serum were measured at different time points: before administration of drugs (T1), at the end of the operation (T2), postoperative 2 hour (T3) and postoperative 24 hour (T4)
Drug: Dexmedetomidine — Participants in the group DEX received dexmedetomidine infusion (0.5 µg/kg loading, 0.4 µg/kg/h infusion) until 30 min before the end of the operation. Interleukin-6 and tumor necrosis factor-α levels in serum were measured at different time points: before administration of drugs (T1), at the end of the operation (T2), postoperative 2 hour (T3) and postoperative 24 hour (T4)
Drug: Lidocaine plus Dexmedetomidine — Participants in the group LIDO+DEX were received lidocaine (1.5 mg/kg loading, 1.5 mg/kg/h infusion) and dexmedetomidine infusion (0.5 μg/kg loading, 0.4 μg/kg/h infusion) until 30 min before the end of the operation, respectively. Interleukin-6 and tumor necrosis factor-α levels in serum were measured at different time points: before administration of drugs (T1), at the end of the operation (T2), postoperative 2 hour (T3) and postoperative 24 hour (T4)

SUMMARY:
Objective: The present study was to evaluate the effects of dexmedetomidine alone, lidocaine alone and their combined infusion on postoperative inflammation cytokines after Laparoscopic hysterectomy.

Methods: Investigators enrolled 160 women with American Society of Anesthesiologists (ASA) physical status I and II, aged 40-65 years, and scheduled for elective laparoscopic hysterectomy with general anesthesia from October 2017 to August 2018. The participants were randomly assigned into four groups(n=40 each group): group CON received normal saline infusion, group LIDO received lidocaine infusion (1.5 mg/kg loading, 1.5 mg/kg/h infusion), group DEX received dexmedetomidine infusion (0.5 µg/kg loading, 0.4 µg/kg/h infusion) and group LIDO+DEX received lidocaine (1.5 mg/kg loading, 1.5 mg/kg/h infusion) and dexmedetomidine infusions (0.5 µg/kg loading, 0.4 µg/kg/h infusion). The four groups received an IV bolus infusion of normal saline, lidocaine, dexmedetomidine and lidocaine combined with dexmedetomidine respectively, over 10 minutes before induction of anesthesia, followed by a continuous IV infusion of normal saline, lidocaine, dexmedetomidine and lidocaine combined with dexmedetomidine until abdominal wound closure, respectively. Interleukin-6 and tumor necrosis factor-α levels in serum were measured at different time points: before administration of drugs (T1), the end of surgery (T2), postoperative 2 hour (T3) and postoperative 24 hour (T4).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* weighted 50 kg-65 kg
* aged 40-65 yr
* elective laparoscopic hysterectomy with general anesthesia

Exclusion Criteria:

* a history of allergy to local anesthetics
* severe respiratory, renal or hepatic disease
* preoperative opioids medication
* psychiatric medical history
* Patients with severe hypotension [mean arterial pressure (MAP<60 mmHg)] or bradycardia [heart rate (HR) <40 beats per minute (bpm)], arrhythmia, or urticaria due to lidocaine and dexmedetomidine infusion during the surgery

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 | postoperative 24 hours
  Interleukin-6 level in serum was measured at the before administration of drugs (T1), Interleukin-6 level in serum was measured at the end of the operation (T2); Interleukin-6 level in serum was measured at the postoperative 2 hour (T3); Interleukin-6 level in serum was measured at the postoperative 24 hour (T4)
Tumor necrosis factor-α | postoperative 24 hours
  Tumor necrosis factor-α level in serum was measured at the before administration of drugs (T1); Tumor necrosis factor-α level in serum was measured at the end of the operation (T2); Tumor necrosis factor-α level in serum was measured at the postoperative 2 hour (T3); Tumor necrosis factor-α level in serum was measured at the postoperative 24 hour (T4)
Interleukin-1 | postoperative 24 hours
  Interleukin-1 level in serum was measured at the before administration of drugs (T1); Interleukin-1 level in serum was measured at the end of the operation (T2); Interleukin-1 level in serum was measured at the postoperative 2 hour (T3); Interleukin-1 level in serum was measured at the postoperative 24 hour (T4)

CONTACTS AND LOCATIONS:
Overall Officials: Wang shenbing, Study Director — Department of Anqing Hospital Anesthesiology; Xiao jingbo, Principal Investigator — Department of Anqing Hospital Anesthesiology
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu S, Hu S, Ju X, Li Y, Li Q, Wang S. Effects of intravenous lidocaine, dexmedetomidine, and their combination on IL-1, IL-6 and TNF-alpha in patients undergoing laparoscopic hysterectomy: a prospective, randomized controlled trial. BMC Anesthesiol. 2021 Jan 6;21(1):3. doi: 10.1186/s12871-020-01219-z. PMID 33407156